CLINICAL TRIAL: NCT02302079
Title: A Phase 2, Double-Masked, Randomized, Active Controlled Study to Evaluate the Efficacy and Safety of ASP8232 in Reducing Central Retinal Thickness in Subjects With Diabetic Macular Edema
Brief Title: A Study to Evaluate ASP8232 in Reducing Central Retinal Thickness in Subjects With Diabetic Macular Edema (DME)
Acronym: VIDI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8232-CL-3001
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus; Diabetic Macular Edema
Keywords: ASP8232; Diabetes Mellitus; ranibizumab; Diabetic Macular Edema
MeSH Terms: conditions — Diabetes Mellitus | interventions — ASP8232; Ranibizumab; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ASP8232 + sham intravitreal (IVT) injections (Experimental): ASP8232 will be given orally once daily and sham injections 3 times with 1 month intervals
  Interventions: Drug: ASP8232; Other: Sham intravitreal (IVT) injection
- ASP8232 + ranibizumab intravitreal (IVT) injections (Experimental): ASP8232 will be given orally once daily and ranibizumab injections 3 times with 1 month intervals
  Interventions: Drug: ASP8232; Drug: ranibizumab
- Placebo + ranibizumab intravitreal (IVT) injections (Active Comparator): Placebo will be given orally once daily and ranibizumab injections 3 times with 1 month intervals
  Interventions: Drug: ranibizumab; Drug: Placebo

INTERVENTIONS:
Drug: ASP8232 — oral capsule
  Arms: ASP8232 + ranibizumab intravitreal (IVT) injections; ASP8232 + sham intravitreal (IVT) injections
Drug: ranibizumab — intravitreal (IVT) injection
  Other Names: Lucentis
  Arms: ASP8232 + ranibizumab intravitreal (IVT) injections; Placebo + ranibizumab intravitreal (IVT) injections
Drug: Placebo — oral capsule
  Arms: Placebo + ranibizumab intravitreal (IVT) injections
Other: Sham intravitreal (IVT) injection — intravitreal (IVT) injection
  Arms: ASP8232 + sham intravitreal (IVT) injections

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of ASP8232 in subjects with diabetic macular edema (DME). This study will evaluate the percent change from baseline in excess central subfield thickness (CST) in the study eye as assessed by spectral domain-optical coherence Tomography (SD-OCT) for ASP8232 monotherapy at Month 3.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a documented diagnosis of type 1 or type 2 diabetes mellitus and a glycosylated hemoglobin A1c (HbA1c) of ≤ 12.0% at Screening
* Subject has definite retinal thickening due to diffuse diabetic macular edema (DME) involving the central macula based on evaluating investigator's clinical evaluation and demonstrated by spectral domain-optical coherence tomography (SD-OCT)
* Subject has central subfield thickness (CST) of at least 375 μm by SD-OCT with presence of intraretinal and/or subretinal fluid at screening visit and at the randomization visit
* Subject has early treatment diabetic retinopathy study (ETDRS) best corrected visual acuity (BCVA) letter score ≤ 73 (Snellen 20/40) and ≥ 24 (Snellen 20/320) at screening visit

Exclusion Criteria:

* Subject's study eye has macular edema considered to be due to a cause other than DME
* Subject's study eye has a decrease in BCVA due to causes other than DME that is likely to be decreasing BCVA by 3 lines or more
* Subject's study eye has significant macular ischemia as shown on angiography
* Subject's study eye has any other ocular disease that may cause substantial reduction in BCVA
* Subject has active peri-ocular or ocular infection
* Subject's study eye has a history of non-infectious uveitis
* Subject's study eye has high myopia (-8 diopter or more correction)
* Subject's study eye has a history of prior pars plana vitrectomy
* Subject's study eye has a history of any ocular surgery within 3 months prior to Day 1
* Subject's study eye has a history of YAG capsulotomy within 3 months prior to Day 1
* Subject's study eye has a history of panretinal scatter photocoagulation (PRP) or focal laser within 3 months prior to Day 1 or anticipated need for PRP during the course of the study through the Week 12 visit
* Subject's study eye has a history of prior IVT, subtenon, or periocular, non-sustained release, steroid therapy within 3 months prior to Day 1
* Subject's study eye has a history of intravitreal sustained release dexamethasone therapy within 6 months prior to Day 1.
* Subject's study eye has a history of intravitreal sustained release fluocinolone within 3 years prior to Day 1.
* Subject's study eye has a history of prior treatment for DME with IVT anti-vascular endothelial growth factor (VEGF) treatment within 8 weeks prior to Day 1
* Subject has a history of prior treatment with any other (than previously listed) approved treatment which is not labeled for DME within 1 year prior to Day 1
* Subject's study eye has high-risk proliferative diabetic retinopathy (PDR)
* Subject has uncontrolled glaucoma
* Subject has media clarity, papillary constriction (i.e., senile miosis), or subject lacks cooperation that would interfere with any study procedures, evaluations or interpretation of data

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2016-08-12 (Actual); Study Completion 2016-08-12 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in excess central subfield thickness (CST) in the study eye as assessed by spectral domain-optical coherence tomography (SD-OCT) at Month 3 | Baseline and Month 3

SECONDARY OUTCOMES:
Absolute change from baseline in CST in the study eye as assessed by SD-OCT at Month 3 | Baseline and Month 3
Change from baseline in early treatment diabetic retinopathy study (ETDRS) best corrected visual acuity (BCVA) score in the study eye at Month 3 | Baseline and Month 3
Absolute and percent change from baseline in excess CST in the study eye as assessed by SD-OCT at Months 1 and 2 | Baseline and Months 1, 2

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Lead, Study Director — Astellas Pharma Europe B.V.
Locations (21):
- United States (21):
  - Site US10021, Phoenix, Arizona
  - Site US10025, Tucson, Arizona
  - Site US10006, Arcadia, California
  - Site US10004, Beverly Hills, California
  - Site US10007, Palm Desert, California
  - Site US10011, Sacramento, California
  - Site US10031, Santa Ana, California
  - Site US10029, Golden, Colorado
  - Site US10016, Miami, Florida
  - Site US10005, Winter Haven, Florida
  - Site US10036, Augusta, Georgia
  - Site US10002, Boston, Massachusetts
  - Site US10001, Omaha, Nebraska
  - Site US10027, Reno, Nevada
  - Site US10012, Nashville, Tennessee
  - Site US10010, Abilene, Texas
  - Site US10015, Austin, Texas
  - Site US10013, Houston, Texas
  - Site US10030, McAllen, Texas
  - Site US10009, San Antonio, Texas
  - Site US10017, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Nguyen QD, Sepah YJ, Berger B, Brown D, Do DV, Garcia-Hernandez A, Patel S, Rahhal FM, Shildkrot Y, Renfurm RW; VIDI Research Group. Primary outcomes of the VIDI study: phase 2, double-masked, randomized, active-controlled study of ASP8232 for diabetic macular edema. Int J Retina Vitreous. 2019 Aug 1;5:28. doi: 10.1186/s40942-019-0178-7. eCollection 2019. PMID 31388454
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=298